CLINICAL TRIAL: NCT03631017
Title: Safety, Biodistribution and Radiation Dosimetry of [18F]PARPi
Brief Title: Imaging With a PET Agent for Detection of Cancers of the Head and Neck
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-247
Record Dates: First submitted 2018-08-11; First posted 2018-08-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer
Keywords: Radiation Dosimetry of [18F]PARPi; PET/CT scans
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: This is an open label, investigator initiated single arm, first in human study of a PARP1/2 imaging agent in patients with head and neck squamous cell carcinomas scheduled to undergo surgery.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: [18 F]-PARPi and PET/CT Scans (Experimental): The intervention of this study is the injection of a microdose (< 10 0 ug) of [18 F]- PARPi followed by 3 PET/CT studies to determine the biodistribution of this imaging agent in normal organs as well as the kinetics of uptake in squamous cell carcinomas of the head and neck.
  Interventions: Drug: [18F]- PARPi; Diagnostic Test: PET/CT Scans
- Phase II: [18 F]-PARPi and PET/CT Scans (Experimental): The intervention of this study is the injection of a microdose (< 10 0 ug) of [18 F]- PARPi followed by 3 PET/CT studies to determine the biodistribution of this imaging agent in normal organs as well as the kinetics of uptake in squamous cell carcinomas of the head and neck.
  Interventions: Drug: [18F]- PARPi; Diagnostic Test: PET/CT Scans

INTERVENTIONS:
Drug: [18F]- PARPi — injection of a microdose (< 100 ug) of [18F]- PARPi
Diagnostic Test: PET/CT Scans — Patients will be injected with approximately 10 mCi of [18F]PARPi and a dynamic PET scan of will be acquired for approximately 30 minutes. A second body PET/CT scan will be started approximately 60 min post injection, and a third PET/CT scan will be started at approximately 120 min post injection. The first (dynamic) and the second (body) PET/CT scan will use "ultra -low dose" CT scan for attenuation correction. The last PET/CT scan will be performed with the investigator's regular clinical low-dose CT settings.

SUMMARY:
The purpose of this study is to test the safety of a study drug called PARPi-FL. This drug has been tested in animals but not yet in people. The purpose of this study is to test if a PARPi-FL scan can be used to take pictures of head and neck cancer. The usual approach to imaging this cancer includes several different imaging scans, including x-rays, CT (computed tomography), MRI (magnetic resonance imaging), and PET (positron emission tomography). These tests take pictures of the cancer.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Age ≥18 years
* ECOG performance status 0 or 1
* Biopsy (histologically or cytologically) proven Squamos Cell Carcinoma
* Oral cavity, oropharynx, or nasopharynx primary site
* At least one tumor lesion on standard of care imaging with a minimum diameter of at least 1.5 cm
* Scheduled to undergo treatment at MSKCC
* Willingness to sign informed consent

Part 2

* Age ≥18 years
* ECOG performance status 0 or 1
* Biopsy (histologically or cytologically) proven Squamous Cell Carcinoma
* Oral cavity,oropharynx, or nasopharynx primary site
* Scheduled to undergo surgery (neck dissection and/ or neck dissection + surgical removal of the primary) at MSK
* Willingness to sign informed consent
* Should have had a standard-of-care [18F]-FDG PET/CT scan before surgery (to minimize the possibility of new alterations developing between the two scans both scans should be acquired within a maximum time difference of one month).

Exclusion Criteria:

* Significantly impaired organ function that may interfere with the excretion and metabolism of the imaging agent. Specifically, patients will be excluded if they meet the following criteria:
* Hematologic

  o Platelets <75K/mcL
* Hepatic

  * Bilirubin >2.0 x ULN (institutional upper limits of normal)
  * AST/ALT >2.5 x ULN
* Renal

  o Creatinine > 2.0 x ULN
* Claustrophobia interfering with PET/CT imaging

  * Known allergy to PEG300
  * Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
severity of adverse events | 2 years
  according to Common Terminology Criteria for Adverse Events (CTCAE 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schöder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/